CLINICAL TRIAL: NCT05660512
Title: A Prospective Single Arm Cohort Study of Intraosseous Basivertebral Nerve Ablation
Brief Title: Intracept Intraosseous Basivertebral Nerve Ablation
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Zack McCormick, Principal Investigator; Associate Professor, University of Utah
Other Study IDs: 130205
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intracept Procedure — Radiofrequency ablation of the basivertebral nerve for the relief of chronic vertebrogenic low back pain

SUMMARY:
This is an independent prospective, noninterventional, observational post-market data collection of the patient-reported effectiveness, ongoing safety and satisfaction outcomes for patients treated with the Intracept Procedure at a single study site.

DETAILED DESCRIPTION:
The Investigator Sponsor will initially approach patients planning to undergo the Intracept Procedure to discuss their interest in learning more about the study. With patient permission, contact information will be forwarded to a third-party research organization which will contact the patient to explain more about the study and to gather Verbal Informed Consent.

Study data will be collected by the University of Utah research staff via 4 telephone study visits under the direction of the Sponsor Investigator. The study research staff will enter the study data directly into a study database and issue the subject stipend after the completion of each study visit.

Data will be analyzed by a statistician under the direction of the Sponsor Investigator for this single-site study.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for intraosseous basivertebral nerve ablation with the Intracept Procedure
* OR Participant had an Intracept Procedure for their low back pain and completed standard of care questionnaires at their procedure appointment.

Exclusion Criteria:

* Not scheduled for an intraosseous basivertebral nerve ablation with the Intracept Procedure
* Intracept procedure for different location other than low back pain

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients at the single study site who are offered an Intracept Procedure are eligible and will be approached to participate in this study. Up to 150 participants who are planning to be treated with the Intracept Procedure will be consented and ultimately, 50 participants with 12 months of follow-up data will be followed.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Change | 3 months
  Validated questionnaire of low back pain related disability. Comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 3 months.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) Change | 12 months
  Mean Improvement in ODI scores from baseline (scale 0 to 100):
  Validated questionnaire of low back pain related disability. Comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 3 months.
Oswestry Disability Index (ODI) Change | 24 months
  Mean improvement in ODI scores from baseline (scale 0 to 100):
  Validated questionnaire of low back pain related disability. Comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 3 months.
Numeric Pain Rating Scale (NPRS) | 3 months
  Mean change in patient-reported low back pain from baseline. The scale is from 0 (no pain) to 10 (worst pain imaginable).
Numeric Pain Rating Scale (NPRS) | 12 months
  Mean change in patient-reported low back pain from baseline. The scale is from 0 (no pain) to 10 (worst pain imaginable).
Numeric Pain Rating Scale (NPRS) | 24 months
  Mean change in patient-reported low back pain from baseline. The scale is from 0 (no pain) to 10 (worst pain imaginable).
Combined Responder Rates (improvement thresholds of ODI ≥ 15 and NPRS ≥ 2) | 3 months
  Percent of responders meeting both thresholds
Combined Responder Rates (improvement thresholds of ODI ≥ 15 and NPRS ≥ 2) | 12 months
  Percent of responders meeting both thresholds
Combined Responder Rates (improvement thresholds of ODI ≥ 15 and NPRS ≥ 2) | 24 months
  Percent of responders meeting both thresholds
PROMIS 29 Change | 3 months
  Mean change in PROMIS-29 from baseline. (PROMIS-29 includes Numeric Rating Score (NRS) and Seven Health Domains. [NRS 0-10 zero being none and 10 the worst. Seven health domains scaled 1-5: physical function (1 unable to do to 5 without any difficulty), fatigue (1 not at all and 5 very much), pain interference (1 not at all and 5 very much), depressive symptoms (1 never and 5 always), anxiety (1 never and 5 always), ability to participate in social roles and activities (1 never and 5 always), and sleep disturbance(1 not at all and 5 very much)])
PROMIS 29 Change | 12 months
  Mean change in PROMIS-29 from baseline. (PROMIS-29 includes Numeric Rating Score (NRS) and Seven Health Domains. [NRS 0-10 zero being none and 10 the worst. Seven health domains scaled 1-5: physical function (1 unable to do to 5 without any difficulty), fatigue (1 not at all and 5 very much), pain interference (1 not at all and 5 very much), depressive symptoms (1 never and 5 always), anxiety (1 never and 5 always), ability to participate in social roles and activities (1 never and 5 always), and sleep disturbance(1 not at all and 5 very much)])
PROMIS 29 Change | 24 months
  Mean change in PROMIS-29 from baseline. (PROMIS-29 includes Numeric Rating Score (NRS) and Seven Health Domains. [NRS 0-10 zero being none and 10 the worst. Seven health domains scaled 1-5: physical function (1 unable to do to 5 without any difficulty), fatigue (1 not at all and 5 very much), pain interference (1 not at all and 5 very much), depressive symptoms (1 never and 5 always), anxiety (1 never and 5 always), ability to participate in social roles and activities (1 never and 5 always), and sleep disturbance(1 not at all and 5 very much)])
Quadrants of % reduction in low back pain from baseline to each follow-up period. | 3 months
  Review of the % of low back pain reduction in participants
Quadrants of % reduction in low back pain from baseline to each follow-up period. | 12 months
  Review of the % of low back pain reduction in participants
Quadrants of % reduction in low back pain from baseline to each follow-up period. | 24 months
  Review of the % of low back pain reduction in participants
Responder rates for Oswestry Disability Index (ODI) | 3 months
  The proportion of subjects who achieve ≥ 15-point reduction in ODI from baseline to each follow-up period. This would indicate a reduction in how much lower back pain is affecting participants' daily activities following the procedure.
  The Oswestry Disability Index (ODI) is a validated questionnaire of low back pain related disability comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 3 months.
Responder rates for Oswestry Disability Index (ODI) | 12 months
  The proportion of subjects who achieve ≥ 15-point reduction in ODI from baseline to each follow-up period. This would indicate a reduction in how much lower back pain is affecting participants' daily activities following the procedure.
  The Oswestry Disability Index (ODI) is a validated questionnaire of low back pain related disability comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 12 months.
Responder rates for Oswestry Disability Index (ODI) | 24 months
  The proportion of subjects who achieve ≥ 15-point reduction in ODI from baseline to each follow-up period. This would indicate a reduction in how much lower back pain is affecting participants' daily activities following the procedure.
  The Oswestry Disability Index (ODI) is a validated questionnaire of low back pain related disability comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 24 months.
Responder rates for the Numeric Pain Rating Scale (NPRS) | 3 Months
  The proportion of subjects who achieve a ≥ 2-point reduction in the NPRS from baseline to each follow-up period. The scale is from 0 (no pain) to 10 (worst pain imaginable).
Responder rates the Numeric Pain Score | 12 Months
  the proportion of subjects who achieve a ≥ 2-point reduction in numeric pain score from baseline to each follow-up period. The scale is from 0 (no pain) to 10 (worst pain imaginable).
Responder rates for the Numeric Pain Score | 24 Months
  the proportion of subjects who achieve a ≥ 2-point reduction in numeric pain score from baseline to each follow-up period. The scale is from 0 (no pain) to 10 (worst pain imaginable).
Narcotic use | 3 Months
  The proportion of patients actively utilizing narcotics for low back pain at each follow-up period.
Narcotic use | 12 Months
  The proportion of patients actively utilizing narcotics for low back pain at each follow-up period.
Narcotic use | 24 Months
  The proportion of patients actively utilizing narcotics for low back pain at each follow-up period.
Low back pain injections | 3 Months
  The proportion of patients utilizing injections for low back pain of the same treatment region at each follow-up period.
Low back pain injections | 12 Months
  The proportion of patients utilizing injections for low back pain of the same treatment region at each follow-up period.
Low back pain injections | 24 Months
  The proportion of patients utilizing injections for low back pain of the same treatment region at each follow-up period.
Low back pain interventions or surgery | 3 Months
  The proportion of patients with pain interventions or surgery for low back pain of the same treatment region at each follow-up period
Low back pain interventions or surgery | 12 Months
  The proportion of patients with pain interventions or surgery for low back pain of the same treatment region at each follow-up period
Low back pain interventions or surgery | 24 Months
  The proportion of patients with pain interventions or surgery for low back pain of the same treatment region at each follow-up period
Work Impact | 12 Months
  Patient work status at 12 months indicated by subject using this scale: No impact to my ability to work; Working with restrictions; Had to get a different job due to low back pain; Unable to work at all/disabled by my low back pain (e.g. retired, unemployed); Not currently working unrelated to low back pain; Other.
  If a subject is working with restrictions, they are asked to specify: Reduced hours; Slower pace; Less heavy work; Not regular job.
  Subjects are also asked the question: How many workdays have you missed due to low back pain?
Patient Global Impression of Change (PGIC) | 3 Months
  PGIC at each follow-up period. The subject is asked to rate their low back pain progress with the scale: Very Much Improved; Much Improved; Minimally Improved; No Change; Minimally worse; Much Worse; Very Much Worse.
Patient Global Impression of Change (PGIC) | 12 Months
  PGIC at each follow-up period. The subject is asked to rate their low back pain progress with the scale: Very Much Improved; Much Improved; Minimally Improved; No Change; Minimally worse; Much Worse; Very Much Worse.
Patient Global Impression of Change (PGIC) | 24 Months
  PGIC at each follow-up period. The subject is asked to rate their low back pain progress with the scale: Very Much Improved; Much Improved; Minimally Improved; No Change; Minimally worse; Much Worse; Very Much Worse.
Patient-reported procedure-related adverse events | 3 Months
  Patient-reported procedure-related adverse events including new LBP and/or leg pain at each follow-up period
Patient-reported procedure-related adverse events | 12 Months
  Patient-reported procedure-related adverse events including new LBP and/or leg pain at each follow-up period
Patient-reported procedure-related adverse events | 24 Months
  Patient-reported procedure-related adverse events including new LBP and/or leg pain at each follow-up period

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Utah Farmington Health Center, Farmington, Utah
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - University of Utah South Jordan Health Center, South Jordan, Utah

REFERENCES:
- [Background] Lotz JC, Fields AJ, Liebenberg EC. The role of the vertebral end plate in low back pain. Global Spine J. 2013 Jun;3(3):153-64. doi: 10.1055/s-0033-1347298. Epub 2013 May 23. PMID 24436866
- [Background] Dudli S, Fields AJ, Samartzis D, Karppinen J, Lotz JC. Pathobiology of Modic changes. Eur Spine J. 2016 Nov;25(11):3723-3734. doi: 10.1007/s00586-016-4459-7. Epub 2016 Feb 25. PMID 26914098
- [Background] Munir S, Freidin MB, Rade M, Maatta J, Livshits G, Williams FMK. Endplate Defect Is Heritable, Associated With Low Back Pain and Triggers Intervertebral Disc Degeneration: A Longitudinal Study From TwinsUK. Spine (Phila Pa 1976). 2018 Nov 1;43(21):1496-1501. doi: 10.1097/BRS.0000000000002721. PMID 29847371
- [Background] Dudli S, Sing DC, Hu SS, Berven SH, Burch S, Deviren V, Cheng I, Tay BKB, Alamin TF, Ith MAM, Pietras EM, Lotz JC. ISSLS PRIZE IN BASIC SCIENCE 2017: Intervertebral disc/bone marrow cross-talk with Modic changes. Eur Spine J. 2017 May;26(5):1362-1373. doi: 10.1007/s00586-017-4955-4. Epub 2017 Jan 31. PMID 28138783
- [Background] Fras C, Kravetz P, Mody DR, Heggeness MH. Substance P-containing nerves within the human vertebral body. an immunohistochemical study of the basivertebral nerve. Spine J. 2003 Jan-Feb;3(1):63-7. doi: 10.1016/s1529-9430(02)00455-2. PMID 14589248
- [Background] Bailey JF, Liebenberg E, Degmetich S, Lotz JC. Innervation patterns of PGP 9.5-positive nerve fibers within the human lumbar vertebra. J Anat. 2011 Mar;218(3):263-70. doi: 10.1111/j.1469-7580.2010.01332.x. Epub 2011 Jan 12. PMID 21223256
- [Background] Fischgrund JS, Rhyne A, Franke J, Sasso R, Kitchel S, Bae H, Yeung C, Truumees E, Schaufele M, Yuan P, Vajkoczy P, DePalma M, Anderson DG, Thibodeau L, Meyer B. Intraosseous basivertebral nerve ablation for the treatment of chronic low back pain: a prospective randomized double-blind sham-controlled multi-center study. Eur Spine J. 2018 May;27(5):1146-1156. doi: 10.1007/s00586-018-5496-1. Epub 2018 Feb 8. PMID 29423885
- [Background] Fischgrund JS, Rhyne A, Franke J, Sasso R, Kitchel S, Bae H, Yeung C, Truumees E, Schaufele M, Yuan P, Vajkoczy P, Depalma M, Anderson DG, Thibodeau L, Meyer B. Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain: 2-Year Results From a Prospective Randomized Double-Blind Sham-Controlled Multicenter Study. Int J Spine Surg. 2019 Apr 30;13(2):110-119. doi: 10.14444/6015. eCollection 2019 Apr. PMID 31131209
- [Background] Fischgrund JS, Rhyne A, Macadaeg K, Moore G, Kamrava E, Yeung C, Truumees E, Schaufele M, Yuan P, DePalma M, Anderson DG, Buxton D, Reynolds J, Sikorsky M. Long-term outcomes following intraosseous basivertebral nerve ablation for the treatment of chronic low back pain: 5-year treatment arm results from a prospective randomized double-blind sham-controlled multi-center study. Eur Spine J. 2020 Aug;29(8):1925-1934. doi: 10.1007/s00586-020-06448-x. Epub 2020 May 25. PMID 32451777
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727
- [Background] Hagg O, Fritzell P, Nordwall A; Swedish Lumbar Spine Study Group. The clinical importance of changes in outcome scores after treatment for chronic low back pain. Eur Spine J. 2003 Feb;12(1):12-20. doi: 10.1007/s00586-002-0464-0. Epub 2002 Oct 24. PMID 12592542
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Ostelo RW, de Vet HC. Clinically important outcomes in low back pain. Best Pract Res Clin Rheumatol. 2005 Aug;19(4):593-607. doi: 10.1016/j.berh.2005.03.003. PMID 15949778